CLINICAL TRIAL: NCT06567496
Title: The Effects of a Virtual Reality Intervention on Mental Health Outcomes and Academic Success in First Year Physical Therapy Students
Brief Title: Effects of a Virtual Reality Intervention on Mental Health Outcomes and Academic Success in Physical Therapy Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Belmont University (Other)
Collaborators: BehaVR LLC (Industry)
Responsible Party: Principal Investigator, Sue Curfman, Associate Professor, Belmont University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BelmontU
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Mental Stress; Anxiety; Depression; Satisfaction
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Mixed methods randomized controlled trial with a waitlist control group incorporating focus groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 8 week First Resort virtual reality navigated through Meta Quest II headset devices
  Interventions: Other: First Resort
- Delayed experimental intervention group (Other): 8 week First Resort virtual reality navigated through Meta Quest II headset devices delayed by one semester
  Interventions: Other: First Resort

INTERVENTIONS:
Other: First Resort — First Resort is an 8-week, self-guided, at-home, virtual reality program designed to be navigated via Meta Quest II headset devices and will be used as an intervention.
  Other Names: First

SUMMARY:
Exploring the impact of a virtual reality program, First Resort on graduate physical therapy student wellness and academic success.

DETAILED DESCRIPTION:
This study is exploring the impact of an 8-week virtual reality intervention among graduate physical therapy students. Self-report measures of anxiety, depression and stress will be collected pre/post to assess the impact of the virtual reality intervention.

Purpose:

1. Determine if there is an impact of a virtual reality intervention on symptoms of anxiety, depression and stress levels in first year physical therapy doctoral students
2. Explore correlations between performance, anxiety, depression, stress and First Resort use in first year physical therapy doctoral students
3. Explore the feasibility of use of First Resort app in first year physical therapy doctoral students

ELIGIBILITY:
Inclusion Criteria:

Physical Therapy students enrolled at a single university in the southern United States during the fall 2024 semester

-

Exclusion Criteria:

Patient Health Questionnaire-8 score of 15 or more General Anxiety Disorder-7 score of 15 or more History of seizures History of motion sickness History of epilepsy History of balance impairment History of significant visual History of auditory impairment

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 | 8 weeks
  Self-reported questionnaire most frequently used worldwide for the screening and severity assessment of depression. Minimum score of 0 indicating no or minimal depression and maximum of 24 which is severe depression.
General Anxiety Disorder-7 | 8 weeks
  Self-reported questionnaire to measure or assess the severity of generalized anxiety disorder. Minimum score of 0 indicating no or minimal anxiety and maximum of 21 which is severe anxiety.
Perceived Stress Scale-10 | 8 weeks
  Self-reported measure of global perceived stress. Minimum score of 0 indicating low perceived stress and maximum of 40 which high perceived stress.
Client Satisfaction Questionnaire-8 | 8 weeks
  Self-reported questionnaire assessing satisfaction with the intervention. Minimum score of 8 indicating low satisfaction and maximum of 32 which is very high satisfaction.
Self-reported Cumulative Grade Point Average | 8 weeks
  Participants self-report the overall semester grade point average. 0.0-4.0 with 0.0 indicating failure and 4.0 indicating all A's.

SECONDARY OUTCOMES:
Patient Health Questionnaire-2 | 8 weeks
  Self-reported questionnaire most frequently used worldwide for the screening and severity assessment of depression. Minimum score 0 indicating low likelihood depression and maximum of 6 which indicates positive screen for depression.
General Anxiety Disorder-2 | 8 weeks
  Self-reported questionnaire to measure or assess the severity of generalized anxiety disorder. Minimum score 0 indicating low likelihood of anxiety and maximum of 6 which indicates positive screen for anxiety.
The exit survey included several questions about Life style factors | 8 weeks
  Participants will be asked about sleep and exercise behaviors throughout the study. They will also be asked if they had mental health support during the study, such as counseling or psychiatric care.
Qualitative feedback_Focus groups | 8 weeks
  Describe experience with study through open-ended questions informing discussion portion of the paper.
Descriptive categorical | 8 weeks
  This is descriptive and categorical data delivered through Qualtrics using single choice from multiple categorical responses. This included descriptive information about sleep, exercise habits, and other consults sought by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sue E Curfman, PT, DHSc, Principal Investigator — Belmont University
Locations (1):
- Belmont University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoying J, Melnyk BM, Hutson E, Tan A. Prevalence and Correlates of Depression, Anxiety, Stress, Healthy Beliefs, and Lifestyle Behaviors in First-Year Graduate Health Sciences Students. Worldviews Evid Based Nurs. 2020 Feb;17(1):49-59. doi: 10.1111/wvn.12415. Epub 2020 Jan 8. PMID 31912989
- [Background] Bolinski F, Etzelmuller A, De Witte NAJ, van Beurden C, Debard G, Bonroy B, Cuijpers P, Riper H, Kleiboer A. Physiological and self-reported arousal in virtual reality versus face-to-face emotional activation and cognitive restructuring in university students: A crossover experimental study using wearable monitoring. Behav Res Ther. 2021 Jul;142:103877. doi: 10.1016/j.brat.2021.103877. Epub 2021 May 11. PMID 34029860
- [Background] Ma J, Zhao D, Xu N, Yang J. The effectiveness of immersive virtual reality (VR) based mindfulness training on improvement mental-health in adults: A narrative systematic review. Explore (NY). 2023 May-Jun;19(3):310-318. doi: 10.1016/j.explore.2022.08.001. Epub 2022 Aug 5. PMID 36002363
- [Background] Macauley K, Plummer L. Prevalence and Predictors of Anxiety in Doctor of Physical Therapy Students. J Allied Health. 2017 Summer;46(2):e39-e41. PMID 28561872
- See also: A mental wellness game for Quest Virtual Reality. First Resort. (2022, November 28). — https://www.realizedcare.com/stress
- See also: Stress, worry & sadness. RealizedCare — http://www.realizedcare.com/stress